CLINICAL TRIAL: NCT02703662
Title: Performance of Biologic Mesh Materials in Abdominal Wall Reconstruction - A Randomized Controlled Trial
Brief Title: Performance of Biologic Mesh Materials in Abdominal Wall Reconstruction
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Calgary (Other)
Collaborators: Medtronic (Industry)
Responsible Party: Principal Investigator, Dr. Chad G. Ball, Associate Professor, University of Calgary
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Bio_ Mesh
Record Dates: First submitted 2016-02-25; First posted 2016-03-09 (Estimated); Last update posted 2023-02-03 (Actual); Status verified 2023-02

CONDITIONS: Ventral Hernia
Keywords: Biologic mesh; abdominal wall reconstruction
MeSH Terms: conditions — Hernia, Ventral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Strattice biologic mesh (Active Comparator): Strattice mesh is made of noncross-linked porcine dermis, which is used to support abdominal wall reconstruction.
  Interventions: Device: Strattice biologic mesh
- Permacol biologic mesh (Experimental): Permacol mesh is made of cross-linked porcine dermis, which is used to support abdominal wall reconstruction.
  Interventions: Device: Permacol biologic mesh

INTERVENTIONS:
Device: Strattice biologic mesh — Patients randomized to this group will be inserted one or more Strattice biologic meshes during the abdominal wall reconstruction surgical procedure.
  Arms: Strattice biologic mesh
Device: Permacol biologic mesh — Patients randomized to this group will be inserted one or more Permacol biologic meshes during the abdominal wall reconstruction surgical procedure.
  Arms: Permacol biologic mesh

SUMMARY:
To date, there have been no prospective randomized controlled trials that compare various biologic mesh materials in the context of abdominal wall reconstruction. As a result, this proposal describes a 'head to head' randomized controlled trial (RCT) between 2 of the market's most popular biologic meshes. Strattice (noncross-linked porcine dermis, LifeCell Inc.) will be compared to Permacol (cross-linked porcine dermis, Covidien Inc.) in a randomized manner. Although there are significant differences between these mesh products with regard to procurement, tissue processing and cost, clinical controlled trials are needed to compare their performance.

DETAILED DESCRIPTION:
Complex abdominal wall reconstructions utilize advanced techniques that include, but are not limited to, component separation, modified component separation, and free tissue flap reconstruction. Data suggests that recurrence rates are lowered with the insertion of mesh supporting materials. More specifically, synthetic mesh utilization during repair of simple clean ventral hernias reduces hernia recurrence by over 50% when compared to suture closure alone. Unfortunately in the presence of microbial contamination or infection, there is a marked increase in hernia recurrence and mesh infection using synthetic prostheses. Biologic meshes however are established options for use in abdominal wall reconstruction in the presence of both field contamination and infection. These indications, as well as others, for biologic materials include, but are not limited to, patients with chronic immunosuppression, infected fields, colonized fields (i.e. preceding synthetic mesh), the need to place the product within the peritoneal cavity (underlay), and patients with complex losses of domain. It should also be noted that there may be significant utility in their use of biologic materials in a much broader range of indications, but the economic cost of these products have clearly tempored wider indications for overall use.

To date, there have been no prospective randomized controlled trials that compare various biologic mesh materials in the context of abdominal wall reconstruction. As a result, this proposal describes a 'head to head' randomized controlled trial (RCT) between 2 of the market's most popular biologic meshes. Strattice (noncross-linked porcine dermis, LifeCell Inc.) will be compared to Permacol (cross-linked porcine dermis, Covidien Inc.) in a randomized manner. Although there are significant differences between these mesh products with regard to procurement, tissue processing and cost, clinical controlled trials are needed to compare their performance.

Given the nearly 2-fold difference in cost between the 2 included biologic meshes, equivalence with regard to recurrence and postoperative complications would represent a massive economic savings to the public health care system.

ELIGIBILITY:
Inclusion Criteria:

* The study population will consist of adult patients, 18 years or older, undergoing an abdominal wall reconstruction. Prior to selection, at least 2 surgeons involved in the trial must agree that the indication for use of biologic implant is mutual.

Exclusion Criteria:

* Patients will be excluded if they are unable or unwilling to provide informed consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2017-10-26 (Actual); Primary Completion 2025-10 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
The percentage of hernia recurrence in patients received the biologic meshes. | 12 months postoperation

SECONDARY OUTCOMES:
The percentage of wound infection of the participants. | 12 months postoperation
The days of hospital stay post the abdominal wall reconstruction procedure. | 12 months postoperation

CONTACTS AND LOCATIONS:
Locations (1):
- Foothills Medical Centre, Faculty of Medicine, Calgary, Alberta, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Burger JW, Luijendijk RW, Hop WC, Halm JA, Verdaasdonk EG, Jeekel J. Long-term follow-up of a randomized controlled trial of suture versus mesh repair of incisional hernia. Ann Surg. 2004 Oct;240(4):578-83; discussion 583-5. doi: 10.1097/01.sla.0000141193.08524.e7. PMID 15383785
- [Background] Richmond BK, Chong B. Routine use of bioprosthetic mesh is not necessary: a retrospective review of 100 consecutive cases of intra-abdominal midweight polypropylene mesh for ventral hernia repair. Surgery. 2013 May;153(5):741. doi: 10.1016/j.surg.2013.02.006. Epub 2013 Mar 13. No abstract available. PMID 23489939
- [Background] Leber GE, Garb JL, Alexander AI, Reed WP. Long-term complications associated with prosthetic repair of incisional hernias. Arch Surg. 1998 Apr;133(4):378-82. doi: 10.1001/archsurg.133.4.378. PMID 9565117
- [Background] Rosen MJ, Krpata DM, Ermlich B, Blatnik JA. A 5-year clinical experience with single-staged repairs of infected and contaminated abdominal wall defects utilizing biologic mesh. Ann Surg. 2013 Jun;257(6):991-6. doi: 10.1097/SLA.0b013e3182849871. PMID 23426340
- [Background] Lupinacci RM, Gizard AS, Rivkine E, Debove C, Menegaux F, Barrat C, Wind P, Tresallet C. Use of a bioprosthetic mesh in complex hernia repair: early results from a French multicenter pilot study. Surg Innov. 2014 Dec;21(6):600-4. doi: 10.1177/1553350613520514. Epub 2014 Feb 3. PMID 24496103
- [Background] Iacco A, Adeyemo A, Riggs T, Janczyk R. Single institutional experience using biological mesh for abdominal wall reconstruction. Am J Surg. 2014 Sep;208(3):480-4; discussion 483-4. doi: 10.1016/j.amjsurg.2013.09.020. Epub 2013 Dec 25. PMID 24462172
- [Background] Ouellet JF, Ball CG, Kortbeek JB, Mack LA, Kirkpatrick AW. Bioprosthetic mesh use for the problematic thoracoabdominal wall: outcomes in relation to contamination and infection. Am J Surg. 2012 May;203(5):594-597. doi: 10.1016/j.amjsurg.2012.01.008. Epub 2012 Mar 23. PMID 22444712
- [Background] Kirkpatrick AW, Roberts DJ, De Waele J, Jaeschke R, Malbrain ML, De Keulenaer B, Duchesne J, Bjorck M, Leppaniemi A, Ejike JC, Sugrue M, Cheatham M, Ivatury R, Ball CG, Reintam Blaser A, Regli A, Balogh ZJ, D'Amours S, Debergh D, Kaplan M, Kimball E, Olvera C; Pediatric Guidelines Sub-Committee for the World Society of the Abdominal Compartment Syndrome. Intra-abdominal hypertension and the abdominal compartment syndrome: updated consensus definitions and clinical practice guidelines from the World Society of the Abdominal Compartment Syndrome. Intensive Care Med. 2013 Jul;39(7):1190-206. doi: 10.1007/s00134-013-2906-z. Epub 2013 May 15. PMID 23673399
- [Background] Bellows CF, Smith A, Malsbury J, Helton WS. Repair of incisional hernias with biological prosthesis: a systematic review of current evidence. Am J Surg. 2013 Jan;205(1):85-101. doi: 10.1016/j.amjsurg.2012.02.019. Epub 2012 Aug 4. PMID 22867726
- [Background] Smart NJ, Marshall M, Daniels IR. Biological meshes: a review of their use in abdominal wall hernia repairs. Surgeon. 2012 Jun;10(3):159-71. doi: 10.1016/j.surge.2012.02.006. Epub 2012 Mar 20. PMID 22436406
- [Background] Cheng AW, Abbas MA, Tejirian T. Outcome of abdominal wall hernia repair with biologic mesh: Permacol versus Strattice. Am Surg. 2014 Oct;80(10):999-1002. PMID 25264647
- [Background] Melnik I, Goldstein D, Yoffe B. Use of a porcine dermal collagen implant for contaminated abdominal wall reconstruction in a 105-year-old woman: a case report and review of the literature. J Med Case Rep. 2015 Apr 29;9:95. doi: 10.1186/s13256-015-0569-9. PMID 25925149
- [Derived] Carver DA, Kirkpatrick AW, Eberle TL, Ball CG. Performance of biological mesh materials in abdominal wall reconstruction: study protocol for a randomised controlled trial. BMJ Open. 2019 Feb 15;9(2):e024091. doi: 10.1136/bmjopen-2018-024091. PMID 30772851